CLINICAL TRIAL: NCT04115618
Title: Simultaneous Integrated Boost Intensity-modulated Chemoradiotherapy in Upper Thoracic Esophageal Squamous Cell Carcinoma: a Phase II Study of Single Institution
Brief Title: SIB in Upper Thoracic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-ESCCSIB
Record Dates: First submitted 2019-09-29; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal cancer; Chemoradiotherapy; Simultaneous Integrated Boost Intensity
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: Using IMRT technology, two fields are irradiated synchronously, prescription radiation dose: 50.4 Gy/28F in PTV-C, 1.8 Gy per fraction; 63 Gy/28F in PTV-G, 2.25 Gy per fraction. Six times of concurrent DP week regimen chemotherapy: cisplatin 20mg/m2 qw plus docetaxel 20mg/m2 qw.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIB (Experimental): Simultaneous integrated boost intensity-modulated chemoradiotherapy
  Interventions: Radiation: Simultaneous integrated boost intensity-modulated chemoradiotherapy

INTERVENTIONS:
Radiation: Simultaneous integrated boost intensity-modulated chemoradiotherapy — Using IMRT technology, two fields are irradiated synchronously, prescription radiation dose: 50.4 Gy/28F in PTV-C, 1.8 Gy per fraction; 63 Gy/28F in PTV-G, 2.25 Gy per fraction. Six times of concurrent DP week regimen chemotherapy: cisplatin 20mg/m2 qw plus docetaxel 20mg/m2 qw.

SUMMARY:
This study was designed to predict the toxicity and efficacy of Simultaneous Integrated Boost Intensity-modulated Chemoradiotherapy in Upper Thoracic I-IVA Esophageal Squamous Cell Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytologic diagnosis of esophageal squamous carcinoma;
2. Aged 18-75 years;
3. KPS ≥ 70;
4. Upper thoracic esophageal squamous carcinoma: the upper margin of the lesion is located between the entrance of esophagus and the inferior edge of the azygos vein;
5. Stage I-IVA(AJCC 6th,2009);
6. Not able to be surgically resection or rejected;
7. Not have received any prior anticancer therapy;
8. No serious system dysfunction and immuno-deficiency, Adequate organ function including the following: Hemoglobin ≥9 g/dL, WBC≥4x109/L, Neutrophils (ANC )≥1.5x10^9/L, platelet count ≥100x 10^9/L, serum creatinine<1.5 mg/dL,urea nitrogen <8 mmol/L;
9. No history of malignancy;
10. No perforation of esophagus, no deep ulcer of esophagus;
11. Joined the study voluntarily and signed informed consent form.

Exclusion Criteria:

1. Pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives;
2. Patient who has metastasis such as lung, liver metastasis;
3. Other malignant tumors;
4. Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior;
5. Uncontrollable heart disease, diabetes and hypertension, pulmonary fibrosis, and chest confirmed active pulmonary inflammation require antibiotic treatment, as well as superior vena cava compression syndrome;
6. After surgery, exploratory thoracotomy, radiotherapy, chemotherapy, or targeting therapy;
7. Combination of pure red cell anemia or gamma globulin;
8. Allergic to any medication component studied.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity Effect | 8 Weeks
  Toxicity effect defined as over CTCAE 4 grade 3 acute radiation toxicity of esophagitis 2 weeks after completion of 6 weeks of radiation therapy.

SECONDARY OUTCOMES:
PFS | One month
  Time of disease progression or unrecorded time of death due to any cause from the day of admission to the first imaging confirmation
OS | One month
  Time from admission to death

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No